CLINICAL TRIAL: NCT05932901
Title: A Multinational, Observational, Secondary Data Study Describing Management and Treatment With Dapagliflozin in Routine Clinical Practice Among Patients With Chronic Kidney Disease
Brief Title: OPTIMISE-CKD Drug Utilization
Acronym: OPTIMISE-CKD
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D169AR00015
Record Dates: First submitted 2023-05-05; First posted 2023-07-06 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Dapagliflozin 10mg initiators: Adult patients (aged ≥18 years) with chronic kidney disease, who received a dapagliflozin 10mg prescription on or after the country-specific CKD indication approval date, and who did not previously have a prescription for dapagliflozin.
- Dapagliflozin 10mg eligible but untreated: Adult patients (aged ≥18 years) with chronic kidney disease, who meet the country-specific approved dapagliflozin 10mg treatment criteria for CKD on or after the local CKD indication approval date, but have not received a prescription
- Incident CKD: Adults patients (aged ≥18 years) who newly meet the CKD definition (diagnosis or laboratory indication) during the study period.

SUMMARY:
This is a multi-national, observational study program using secondary data sources to address research questions related to 1) real-world dapagliflozin utilisation in CKD and potential for further utilisation, 2), the current CKD treatment landscape and 3) real-world effectiveness of dapagliflozin in CKD (pending feasibility assessment).

DETAILED DESCRIPTION:
OPTIMISE-CKD is an observational study program using secondary data sources to address research questions related to 1) real-world dapagliflozin utilisation in CKD and potential for further utilisation, 2), the current CKD treatment landscape and 3) real-world effectiveness of dapagliflozin in CKD (pending feasibility assessment).

Primary objective: to characterize dapagliflozin 10mg utilisation in clinical practice, by describing treatment naïve patients who (1) are treated with dapagliflozin 10 mg and (2) who are eligible for CKD treatment with dapagliflozin but untreated.

Secondary objectives: to describe the current clinical landscape among incident CKD patients, by:

1. Describing baseline demographic and clinical characteristics, drug utilization, and CKD treatment (RAASi and dapagliflozin 10 mg) patterns; and
2. Describing selected outcomes among overall, treated and untreated incident CKD patients.

Exploratory objectives: to assess the real-world effectiveness of dapagliflozin in CKD patients, pending feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged ≥18 years)
* Chronic kidney disease (diagnosis code, uACR >30mg/g or 2 eGFR ≥90 days apart, second value ≥75ml/min/1.73m2)
* ≥365 days continuous enrolment in database

Exclusion Criteria:

* History of type 1 diabetes, gestational diabetes or dialysis
* History of dapagliflozin 10mg prescriptions before index date

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The overall study population will consist of adult (aged > 18 years) patients with CKD
Sampling Method: Non-Probability Sample
Enrollment: 2682052 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Baseline demographics | 1 year pre-index
  Patient demographic characteristics including age, sex, race and insurance type (if data are available)
Baseline clinical characteristics | 1 year pre-index
  Number and proportion of patients with comorbidities, including heart failure, cardiovascular disease, type 2 diabetes, hypertension, hyperkalemia, myocardial infarction, stroke
Baseline comedications | 1 year pre-index
  Number and proportion of patients with comedications for cardiovascular disease, diabetes, hyperkalemia
Baseline eGFR in ml/min/1.73m2 | 1 year pre-index
  Number and proportion of patients with available data mean, standard deviation, median, interquartile range, minimum, maximum
Baseline uACR in mg/g | 1 year pre-index
  Number and proportion of patients with available data mean, standard deviation, median, interquartile range, minimum, maximum
Baseline serum creatinine in mg/dl | 1 year pre-index
  Number and proportion of patients with available data mean, standard deviation, median, interquartile range, minimum, maximum
Baseline calcium in mg/dl | 1 year pre-index
  Number and proportion of patients with available data mean, standard deviation, median, interquartile range, minimum, maximum
Baseline sodium in mmol/L | 1 year pre-index
  Number and proportion of patients with available data mean, standard deviation, median, interquartile range, minimum, maximum
Baseline hemoglobin A1c in % | 1 year pre-index
  Number and proportion of patients with available data Mean, standard deviation, median, interquartile range, minimum, maximum
Baseline hematocrit in % | 1 year pre-index
  Number and proportion of patients with available data Mean, standard deviation, median, interquartile range, minimum, maximum, % patients with value <40
Baseline systolic blood pressure in mmHg | 1 year pre-index
  Number and proportion of patients with available data Mean, standard deviation, median, interquartile range, minimum, maximum

SECONDARY OUTCOMES:
Proportion of patients who initiate cardiorenal protective medication | 1 year post-index
  Treatment initiation (RASi and/or SGLT2i/dapagliflozin 10mg) following incident CKD index date
Proportion of patients who continue cardiorenal protective medication | 1 year post-index
  Treatment persistence (RASi and/or SGLT2i/dapagliflozin 10mg) following initiation after incident CKD index date
Proportion of patients with hospitalisations following incident CKD index | 1 year post-index
  Hospitalisations (any reason, CKD, heart failure) following incident CKD index
Average healthcare cost for specific outcomes/reasons | 1 year post-index
  Healthcare costs related to hospitalisation for CKD, heart failure, atherosclerotic CVD following incident CKD index

CONTACTS AND LOCATIONS:
Locations (4):
- Research Site, Minneota, Minnesota, United States
- Japan (2):
  - Research Site, Kyoto, Kyoto
  - Research Site, Tokyo
- Research Site, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure."Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D169AR00015&attachmentIdentifier=c7c8c97f-9df3-4479-afc8-6716a6fd32ee&fileName=Redacted_CSR_Synopsis.pdf&versionIdentifier=